CLINICAL TRIAL: NCT04157101
Title: Health Coaching for Chronic Multi-symptom Illness
Brief Title: Health Coaching for Chronic Multisymptom Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F3254-R
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pain Predominant Chronic Multisymptom Illness
Keywords: Pain; Veteran; Health Coaching; Clinical Trial; Supportive Psychotherapy; Illness beliefs
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Clinical Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator, assessor, biostatistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health Coaching (Experimental): The 12-session remote health coaching intervention assists Veterans in developing and maintaining health behaviors that meet their life goals. Veterans begin by discussing their symptoms, the impact of their symptoms, and their beliefs about Pain-CMI. Next, the Veteran identifies discrepancies between where they are and where they want to be for 5 lifestyle factors. The first half of treatment focuses on providing education about the 5 lifestyle factors. Veterans are introduced to behavior change/health coaching principles. The major focus is on behavior change and development of long-term healthy habits. During the last session, Veterans develop a long-term plan to maintain behavioral changes after the 12-week program and identify the skills that they can utilize moving forward.
  Interventions: Behavioral: Health Coaching
- Supportive Psychotherapy (Placebo Comparator): Our control will be supportive psychotherapy which will focus on discussing weekly stressors in a supportive, non-directive way. Session content is patient-driven, and sessions focus on emphasizing the patients' strengths, following patients' emotional affect, and building a therapeutic alliance. Participants will be asked to generate the topic they would like to discuss for the session and will complete a worksheet between sessions noting emotional events throughout their week ("A time when I felt stressed was ." ) in order to help identify experiences for discussion in session. The control consists of 12 weekly sessions delivered via telephone or video and will be delivered by bachelor's, or master's level providers.
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Health Coaching — The 12-session remote health coaching intervention assists Veterans in developing and maintaining health behaviors that meet their life goals. Veterans begin by discussing their symptoms, the impact of their symptoms, and their beliefs about Pain-CMI. Next, the Veteran identifies discrepancies between where they are and where they want to be for 5 lifestyle factors. The first half of treatment focuses on providing education about the 5 lifestyle factors. Veterans are introduced to behavior change/health coaching principles. The major focus is on behavior change and development of long-term healthy habits. During the last session, Veterans develop a long-term plan to maintain behavioral changes after the 12-week program and identify the skills that they can utilize moving forward.
  Arms: Health Coaching
Behavioral: Supportive Psychotherapy — Our control will be supportive psychotherapy which will focus on discussing weekly stressors in a supportive, non-directive way. Session content is patient-driven, and sessions focus on emphasizing the patients' strengths, following patients' emotional affect, and building a therapeutic alliance. Participants will be asked to generate the topic they would like to discuss for the session and will complete a worksheet between sessions noting emotional events throughout their week ("A time when I felt stressed was ." ) in order to help identify experiences for discussion in session. The control consists of 12 weekly sessions delivered via telephone or video and will be delivered by bachelor's, or master's level providers.
  Arms: Supportive Psychotherapy

SUMMARY:
The National Academy of Medicine (NAM) labels chronic pain as one of the most extensive health care issues facing our society with "severe impacts on all aspects of the lives of its sufferers."1 Pain predominant chronic multisymptom illness (Pain-CMI, e.g., fibromyalgia) is a particularly debilitating and presumptive service connected condition for Veterans who deployed to the Gulf region. Health coaching is an appealing potential approach to improve the disability of Pain-CMI because it is personalized to the Veteran's unique goals and beliefs about Pain-CMI and it will be widely available as the VA is rolling out health coaching. The goal of this proposal is to understand if health coaching is also efficacious for a complex pain condition, Pain-CMI.

DETAILED DESCRIPTION:
Purpose:

Chronic pain is one of the most common healthcare issues that Veterans face; it can be very debilitating as well as difficult to treat. Pain Predominant Chronic Multi-symptom Illness (CMI) (e.g., fibromyalgia) is a particularly debilitating and treatment-resistant chronic pain condition and a presumptive service-connected condition for Veterans who deployed to the Gulf region from 1990-2021 (VA Benefits Administration, 2018). There is an urgent need for evidence-based non-pharmaceutical treatments for chronic pain. This study will explore the efficacy of remote-delivered health coaching intervention aimed at modifying lifestyle factors of diet, exercise, social connections, stress, and sleep. The control condition will be supportive psychotherapy.

Study Aims:

Primary Aim 1: Determine if remote-delivered health coaching reduces (H1a) disability and (H2a) pain impairment as compared to remote-delivered supportive psychotherapy for Veterans with Pain-CMI. The investigators will also assess the improvement in (H1b) disability and (H2b) pain impairment at the 24-month follow-up.

Primary Aim 2: Determine if health coaching results in more frequent clinically significant improvement in (H3) disability (20%) and (H4) pain impairment (1 point) as compared to supportive psychotherapy.

Secondary Aim 3: Determine if health coaching reduces (H5) physical symptoms, (H6) catastrophizing, (H7) limiting activity and increases (H8) pain control as compared to supportive psychotherapy.

Exploratory Aim 4: Determine if the reduction in (H9) catastrophizing, (H10) limiting activity and increases in (H11) pain control mediate the relationship between health coaching and reductions in disability and pain impairment.

Study Design:

The current proposal is a randomized clinical trial to determine the efficacy of remote-delivered health coaching in reducing disability and pain impairment for Veterans with Pain-CMI as compared to supportive psychotherapy (n=250). Additionally, the investigators will explore mechanisms of change. Participants will complete four assessments at four different timepoints: baseline, 6-week mid treatment (~6 weeks after baseline), post-treatment (~12 weeks after baseline), and 24-week follow-up (~24 weeks after baseline).

ELIGIBILITY:
Inclusion Criteria:

* Study Population. Participants will consist of 250 Veterans with Pain-CMI
* CMI meets Kansas City (Steele) definition of CMI
* reports wide-spread pain rated at least 4 on a 0 to 10 point pain bothersome scale
* rates their activity limitations at least 3 on a 0 to 10 point scale

Exclusion Criteria:

* life-threatening condition,
* severe cognitive impairment
* psychotic disorder, pregnant
* plans to become pregnant in the next year
* suicidal intent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
World Health Organization Disability Assessment Schedule | Post-treatment (12 weeks)
  World Health Organization Disability Assessment Schedule (WHO-DAS 2.0) measures disability which is due to physical and mental health conditions. The WHO-DAS is a 40-item measure and assesses two underlying constructs: activity limitations and deficits in social integration. The items of the WHODAS have a factor loading on a composite score of 0.82 to 0.98. The WHO-DAS has been found to have high reliability and validity. Consistent with IMMPACT, our primary outcomes include a general measure of disability (WHO-DAS) and a pain specific measure. A 20% improvement will be considered clinically significant. The WHO-DAS is scored on a scale of 0-100 with higher scores = worse disability.
Brief Pain Inventory | post-treatment (12-weeks)
  Brief Pain Inventory (BPI). Pain will be assessed using the BPI. The BPI is a 11-item measure of pain severity and interference. The BPI has been recommended as a core measure of clinical trials due to its reliability, validity and responsiveness to clinical intervention. There are 7-items for the pain interference subscale which are scored from 0-10 with higher = worse pain interference.
World Health Organization Disability Assessment Schedule | follow up (24 week)
  World Health Organization Disability Assessment Schedule (WHO-DAS 2.0) measures disability which is due to physical and mental health conditions. The WHO-DAS is a 40-item measure and assesses two underlying constructs: activity limitations and deficits in social integration. The items of the WHODAS have a factor loading on a composite score of 0.82 to 0.98. The WHO-DAS has been found to have high reliability and validity and is scored from 0-100 with higher = worse disability.
Brief Pain Inventory | follow-up (24 weeks)
  Brief Pain Inventory (BPI). We will compare the % who have a 1 point improvement between arms. Pain will be assessed using the BPI. The BPI is a 11-item measure of pain severity and interference. The BPI has been recommended as a core measure of clinical trials due to its reliability, validity and responsiveness to clinical intervention. We will use the 7-item interference scale which is scored on a scale of 0-10 with higher = worse pain interference.

SECONDARY OUTCOMES:
Patient Health Questionnaire-15 | post-treatment (12-weeks)
  Patient Health Questionnaire (PHQ-15). The PHQ-15 measures physical symptoms and is scored from 0-30 with higher scores = worse symptom burden. The PHQ-15 was validated on a sample of 6,000 and found to be reliable, valid and responsive to change.
Illness Perception Questionnaire-Revised | post-treatment (12-weeks)
  Illness Perception Questionnaire-Revised (IPQ-R).17 Perceived control beliefs will be measured by the IPQ-R. The IPQ-R measures a broad range of illness beliefs, including severity of illness consequences, chronicity, and controllability of illness. The IPQ has been found to be reliable and valid among patients with CMI, predictive of outcomes and responsive to clinical intervention. We will use the control subscale where higher scores = greater perceived control.
Pain Catastrophizing Scale | post-treatment (12-weeks)
  The Pain Catastrophizing Scale (PCS). Catastrophizing will be measured by the PCS. The PCS is a 13-item measure of the degree of pain catastrophizing. The PCS is reliable, valid, predictive of outcomes and responsive to clinical intervention. The PCS is scored on a scale of 0-52 with higher = worse catastrophizing.
Behavioral Response to Illness Questionnaire | post-treatment (12-weeks)
  Behavioral Response to Illness Questionnaire. Limiting behaviors will be assessed with the BRIQ which measures behavioral responses to CMI. The BRIQ has four subscales: limiting behaviors, all or nothing behaviors, practical support and emotional support. The BRIQ is reliable, valid and predicts onset of CMI. We will use the limiting behaviors and all or nothing subscales where higher is more limiting and all or nothing behaviors respectively.
World Health Organization Disability Assessment Schedule | post-treatment (12-weeks)
  World Health Organization Disability Assessment Schedule (WHO-DAS 2.0). We will compare the % who decrease by 20% between arms. The WHO-DAS measures disability which is due to physical and mental health conditions. The WHO-DAS is a 40-item measure and assesses two underlying constructs: activity limitations and deficits in social integration. The items of the WHODAS have a factor loading on a composite score of 0.82 to 0.98. The WHO-DAS has been found to have high reliability and validity and is scored from 0-100 with higher = worse disability.
Brief Pain Inventory | post-treatment (12-weeks)
  Brief Pain Inventory (BPI). We will compare the % who have a 1 point improvement between arms. Pain will be assessed using the BPI. The BPI is a 11-item measure of pain severity and interference. The BPI has been recommended as a core measure of clinical trials due to its reliability, validity and responsiveness to clinical intervention. The BPI interference scale is 7 items scored from 0-10 with higher = greater interference.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marie McAndrew, PhD, Principal Investigator — East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ
Locations (1):
- East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT04157101/ICF_000.pdf